CLINICAL TRIAL: NCT00653562
Title: Single Blind, Multi-center, Post Marketing Clinical Study of Zolpidem (Myslee) in Adolescent Patients With Insomnia - Evaluation With Polysomnography
Brief Title: Zolpidem (Myslee) Post Marketing Study in Adolescent Patients With Insomnia - Evaluation With Polysomnography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 6199-JC-0002
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Insomnia; Sleep Initiation and Maintenance Disorders
Keywords: polysomnography; zolpidem; Sleep disorders; adolescent
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients will receive placebo in one part and zolpidem in the other part
  Interventions: Drug: zolpidem

INTERVENTIONS:
Drug: zolpidem — Oral
  Other Names: Myslee

SUMMARY:
To evaluate the efficacy of zolpidem for adolescent insomniacs with polysomnography

DETAILED DESCRIPTION:
The study consists of two parts. All patients will receive placebo in one part and Zolpidem in the other part in a single blind manner. Efficacy will be measured with polysomnography .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having nonorganic insomnia of nonorganic sleep disorder in ICD10

Exclusion Criteria:

* Patients with schizophrenia or manic-depressive illness
* Patients with insomnia caused by physical diseases
* Patients having a history of hypersensitivity to zolpidem
* Patients with attention-deficit hyperactivity disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sleep latency | 2 days

SECONDARY OUTCOMES:
Total hours of sleep | 2 days
Frequency of intermediate awaking | 2 days
Time of intermediate awaking | 2 days
Patient impression | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Kansai
  - Kantou
  - Kyusyu
  - Tōhoku

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=141